CLINICAL TRIAL: NCT02280993
Title: Phase I/II Feasibility Study Combining Brentuximab Vedotin With Second Line Salvage Chemotherapy (DHAP) in Hodgkin Lymphoma Patients Refractory to First Line Chemotherapy or in First Relapse Who Are Eligible for High Dose Treatment Followed by Autologous Peripheral Blood Stem Cell Transplantation (ASCT)
Brief Title: Phase I/II Feasibility Study Combining Brentuximab Vedotin With Second Line Salvage Chemotherapy (DHAP) in Hodgkin Lymphoma Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marjolein Spiering (Other)
Collaborators: Millennium: The Takeda Oncology Company (Industry)
Responsible Party: Sponsor-Investigator, Marjolein Spiering, MSc, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Transplant BRaVE; NL40688.018.12 (Other: The Central Committee on Research Involving Human Subjects (CCMO)); 2012-003097-45 (EudraCT Number)
Record Dates: First submitted 2014-08-19; First posted 2014-11-03 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Hodgkin Lymphoma; Refractory; Relapse
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — Dexamethasone; Cisplatin; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DHAP-BV (Experimental): Brentuximab Vedotin with DHAP chemotherapy follow by Autologous Peripheral Blood Stem Cell Transplantation
  Interventions: Drug: DHAP; Drug: Brentuximab Vedotin; Other: Autologous Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: DHAP — DHAP
  Other Names: Dexamethasone; AraC; Cisplatin
Drug: Brentuximab Vedotin — Brentuximab Vedotin
  Other Names: Adcetris; SGN-35
Other: Autologous Peripheral Blood Stem Cell Transplantation — Autologous Peripheral Blood Stem Cell Transplantation
  Other Names: ASCT

SUMMARY:
To combine Brentuximab Vedotin with Dexamethasone, AraC and Cisplatin (DHAP) chemotherapy in patients with Hodgkin lymphoma (HL) refractory to first line chemotherapy or in first relapse is expected to induce a significantly higher (metabolic) complete remission (CR) rate prior to consolidation with BEAM, as judged by FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose)-PET negativity. This will be compared with published data on DHAP salvage only. Increasing the metabolic CR rate prior to consolidation with high dose chemotherapy and autologous stem cell transplantation (ASCT) is expected to improve progression free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD30+ classical HL (central pathology review; results not required to enroll the patient in the study), primarily refractory to first line chemotherapy or in first relapse after any polychemotherapy regimen (e.g. ABVD (Adriamycin, bleomycin, vinblastine, and dacarbazine), baseline BEACOPP ( bleomycin, etoposide, Adriamycin, cyclophosphamide, Oncovin, procarbazine, and prednisone) or escalated BEACOPP, or other induction regimens)
* In case of relapse, the relapse must be histologically confirmed. In case histology is not possible, at least confirmation of the relapse by fine-needle aspiration is required.
* Measurable disease, as defined in Appendix C i.e. CT scans showing at least 2 or more clearly demarcated lesions with a long axis ≥ 1.5 cm and a short axis diameter ≥ 1.0 cm, or 1 clearly demarcated lesion with a long axis ≥ 2.0 cm and a short axis diameter ≥ 1.0 cm. These lesions must be FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose)-positive
* Age ≥ 18 years (upper age limit for auto stem cell transplantation at the discretion of the participating center)
* WHO ≤ 2 (see appendix A)
* Life expectancy of > 3 months with treatment
* No major organ dysfunction, unless HL-related
* Total bilirubin < 1.5x ULN (unless due to lymphoma involvement of the liver or a known history of Gilbert's syndrome)
* ALT/AST < 3x ULN (unless due to lymphoma involvement of the liver; in that case ALT/AST may be elevated up to 5 x ULN)
* glomerular filtration rate (GFR) > 60 ml/min as estimated by the Cockcroft&Gault formula (appendix D)
* Absolute neutrophil count ≥ 1.5x109/L, unless caused by diffuse bone marrow infiltration by the HL
* Platelets ≥ 100x109/L, unless caused by diffuse bone marrow infiltration by the HL
* Hemoglobin must be >8 g/dL
* Written informed consent
* Able to adhere to the study visit schedule and other protocol requirements
* Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agrees to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
* Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
* Eligible for high dose chemotherapy and autologous peripheral blood stem cell transplantation
* Resolution of toxicities from first-line therapy

Exclusion Criteria:

* Peripheral sensory or motor neuropathy grade ≥ 2
* Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of progressive multifocal leukoencephalopathy
* Symptomatic neurologic disease compromising normal activities of daily living or requiring medications
* Patients who have been using other investigational agents within at least 5 half lives of the most recent agent used prior to enrollment in the study
* Patients who were treated with myelosuppressive chemotherapy or biological therapy ≤ 4 weeks before study inclusion
* Female patients who are both lactating and breast feeding or have a positive serum pregnancy test during the screening period or a positive pregnancy test on Day 1 before first dose of study drug or adults of reproductive potential who are not using effective birth control methods.
* Patients with any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first study drug dose
* Patients who have a history of another primary malignancy less than 3 years before study inclusion or previously diagnosed with another malignancy and have evidence of residual disease, with the exception of non-melanoma skin cancer, completely resected melanoma TNMpT1 and carcinoma in situ of the uterine cervix
* Patients with known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin.
* Patients with known HIV seropositivity, known hepatitis B surface antigen-positivity, or known or suspected active hepatitis C infection
* Patients receiving radiation therapy within 8 weeks prior to start of protocol treatment. Emergency radiation therapy is allowed, as long as measurable disease (at non-irradiated sites) persists.
* Patients with a serious psychiatric disorder that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol

  * Patients who have any severe and/or uncontrolled medical condition or other conditions that could affect their participation in the study such as:Known history of symptomatic congestive heart failure (NYHA III, IV), myocardial infarction ≤ 6 months prior to first study drug
  * Evidence of current serious uncontrolled cardiac arrhythmia, angina pectoris, electrocardiographic evidence of acute ischemia or active conduction system abnormalities
  * Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50%
  * severely impaired pulmonary function as defined as spirometry and DLCO (diffusing capacity of the lung for carbon monoxide) that is 50% or less of the normal predicted value and/or O2 saturation that is 90% or less at rest on room air
  * any active (acute or chronic) or uncontrolled infection/disorders that impair the ability to evaluate the patient or for the patient to complete the study
* nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by this study drug, such as severe hypertension that is not controlled with medical management and thyroid abnormalities when thyroid function cannot be maintained in the normal range by medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
rate of patient with grade 4 Adverse Events | 12 weeks
  The rate of patients with severe toxicity during cycle I-III of the combination treatment (BV + DHAP)

SECONDARY OUTCOMES:
(Severe) Adverse Event | 12 weeks
  (Severe) Adverse Events during the combination treatment

OTHER OUTCOMES:
Response | 12 weeks
  Metabolic CR rate (PET-CT) after the third cycle of BV-DHAP reinduction therapy

CONTACTS AND LOCATIONS:
Overall Officials: Anton Hagenbeek, PhD MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Marie José Kersten, PhD MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Marjolein Spiering, MSc, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (13):
- Rigshospitalet, Copenhagen, Denmark
- France (5):
  - Centre Hospitalier Universitaire, Lille
  - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier et Universitaire, Nantes
  - Hôpital Saint Louis, Paris
  - Institut Gustave Roussy, Paris
- Netherlands (4):
  - Academic Medical Center, Amsterdam
  - Free University Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
- United Kingdom (3):
  - Cambridge University Hospitals NHS Foundation Trust | Addenbrooke's Hospital, Cambridge
  - King's College Hospital NHS Foundation Trust, London
  - Christie Hospital, Manchester, Manchester

REFERENCES:
- [Derived] Driessen J, Zwezerijnen GJC, Schoder H, Kersten MJ, Moskowitz AJ, Moskowitz CH, Eertink JJ, Heymans MW, Boellaard R, Zijlstra JM. Prognostic model using 18F-FDG PET radiomics predicts progression-free survival in relapsed/refractory Hodgkin lymphoma. Blood Adv. 2023 Nov 14;7(21):6732-6743. doi: 10.1182/bloodadvances.2023010404. PMID 37722357
- [Derived] Driessen J, Kersten MJ, Visser L, van den Berg A, Tonino SH, Zijlstra JM, Lugtenburg PJ, Morschhauser F, Hutchings M, Amorim S, Gastinne T, Nijland M, Zwezerijnen GJC, Boellaard R, de Vet HCW, Arens AIJ, Valkema R, Liu RDK, Drees EEE, de Jong D, Plattel WJ, Diepstra A; HOVON Lunenburg Lymphoma Phase I/II Consortium (LLPC). Prognostic value of TARC and quantitative PET parameters in relapsed or refractory Hodgkin lymphoma patients treated with brentuximab vedotin and DHAP. Leukemia. 2022 Dec;36(12):2853-2862. doi: 10.1038/s41375-022-01717-8. Epub 2022 Oct 14. PMID 36241696
- [Derived] Kersten MJ, Driessen J, Zijlstra JM, Plattel WJ, Morschhauser F, Lugtenburg PJ, Brice P, Hutchings M, Gastinne T, Liu R, Burggraaff CN, Nijland M, Tonino SH, Arens AIJ, Valkema R, van Tinteren H, Lopez-Yurda M, Diepstra A, De Jong D, Hagenbeek A. Combining brentuximab vedotin with dexamethasone, high-dose cytarabine and cisplatin as salvage treatment in relapsed or refractory Hodgkin lymphoma: the phase II HOVON/LLPC Transplant BRaVE study. Haematologica. 2021 Apr 1;106(4):1129-1137. doi: 10.3324/haematol.2019.243238. PMID 32273476
- See also: Transplant BRaVE — http://www2.hematologie-amc.nl/TransplantBRaVE_studie